CLINICAL TRIAL: NCT03329066
Title: A Pilot Study to Improve Sleep Quality in Urban High School Students With Asthma
Brief Title: Sleep Quality in High School Students With Asthma - II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jean-Marie Bruzzese, Associate Professor of Applied Developmental Psychology (in Nursing), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAQ9707 - II; 1R21HD086448-01A1 (NIH)
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Asthma; Sleep; Asthma in Children
Keywords: Asthma; Sleep; Adolescents; Urban; Intervention; High school
MeSH Terms: conditions — Asthma | interventions — Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research assistants who interview the teenager and their parents/caregivers will not know to which arm the participants are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MAST - Managing Asthma & Sleep in Teens (Experimental): This is an eight week intervention consisting of 4 group and 4 individual tailored coaching sessions that focuses on both asthma and sleep. In this behavioral medicine intervention, teenagers learn ways to better care for their asthma and sleep hygiene. Teen sessions are delivered in school. Their caregivers will receive four educational booklets that correspond to each group session; topics mirror the objectives of each group and the booklets are sent at the time of each group.
  Interventions: Behavioral: MAST - Managing Asthma & Sleep in Teens
- ASMA - Asthma Self-Management for Adol (Active Comparator): ASMA is an evidence-based intervention for students, caregiver education, and education for students' medical providers. The student intervention consists of 3 group sessions & 5 individual tailored coaching sessions. All sessions are held at school. The caregiver intervention includes 3 educational booklets that correspond to the timing of the student group and 4 brief telephone-counseling sessions to review the booklets, answer questions, and provide strategies to support adolescents' steps to care for their asthma. With caregiver permission, we mail students' healthcare providers a toolkit consisting of (1) a letter informing them their patient is participating in ASMA and is being directed to them for clinical evaluation and (2) summaries of key NHLBI guidelines for treating asthma.
  Interventions: Behavioral: ASMA - Asthma Self-Management for Adol
- Information & Referral Control Group (Placebo Comparator): The information-and-referral control intervention is a student-only intervention that consists of 3 group sessions and 5 individual sessions. Sessions are held once a week at school, where students will receive guideline-based information about asthma and other health topics relevant to adolescents (e.g., nutrition, safety). Students will be referred to their medical providers for asthma and other health concerns; if they do not have a provider, they are given referrals in their community.
  Interventions: Behavioral: Information & Referral Control Group

INTERVENTIONS:
Behavioral: MAST - Managing Asthma & Sleep in Teens — This behavioral intervention will teach teenagers asthma self-care strategies and sleep hygiene.
  Arms: MAST - Managing Asthma & Sleep in Teens
Behavioral: ASMA - Asthma Self-Management for Adol — This behavioral intervention focuses only on asthma care.
  Arms: ASMA - Asthma Self-Management for Adol
Behavioral: Information & Referral Control Group — Students learn basic information about asthma and sleep, as well as other health topics relevant to teenagers.
  Arms: Information & Referral Control Group

SUMMARY:
The overall goal of this project is to develop and to preliminarily validate a novel intervention to be delivered in the high school setting that integrates two evidence-based, school-based interventions for urban adolescents with proven efficacy: (1) Asthma Self-Management for Adolescents (ASMA), an intervention for adolescents with uncontrolled asthma and (2) the Sleep-Smart Program (Sleep-Smart), which focuses on sleep hygiene and behaviors in urban adolescents.

The aim for Phase I is to develop and integrate school-based interventions to improve asthma self-management and sleep hygiene in urban high school students via interviews.

The aims for Phase II are: (1) to evaluate the feasibility and acceptability of the intervention procedures; and (2) to assess the preliminary evidence of the effects of the intervention on improving sleep quality in urban high school students with persistent asthma over a 2-month follow-up period.

This record is for Phase II only.

DETAILED DESCRIPTION:
Sleep quality among adolescents is poor and asthma's impact is significant among adolescents. Asthma control is an important risk factor for poor sleep. In addition, poor asthma control, poor sleep hygiene, and poor sleep quality are more likely in urban settings. Interventions to promote sleep quality by targeting both asthma control and sleep hygiene in this vulnerable population are lacking. We developed a novel intervention -- Managing Asthma and Sleep in Teenagers (MAST) -- and in this phase of the study will evaluate the intervention's feasibility and acceptability and assess the preliminary evidence of intervention effects on improving sleep quality in urban high school students in NYC and Providence, RI. This study is a multi-site trial and collaboration between Columbia University Medical Center and Rhode Island Hospital (RIH).

The investigators hypothesize that: (1) The intervention will be feasible and acceptable as evidenced by adolescents' high rates of adherence to the treatment protocol, and their high satisfaction ratings and positive responses to exit interviews; and (2) relative to controls, over 2-months post-intervention adolescents randomized to the intervention will have significant improvement on the following outcomes assessing sleep quality: (1) sleep efficiency; (2) night awakenings; and (3) sleep duration. If hypotheses are supported, the investigators will explore whether treatment effects on sleep quality outcomes are mediated through changes in asthma self-management (e.g., confidence to care for asthma, steps taken to prevent the onset of symptoms, taking controller medication), and changes in sleep hygiene and behaviors (e.g., consistent bedtime and wake time, consistent sleep location, fewer sleep distractions in child's bedroom, decreased caffeine use). The investigators will also compare MAST to the evidence-based intervention -- Asthma Self-Management for Adolescents (ASMA) -- to explore if whether an asthma intervention integrated with sleep hygiene components enhances sleep quality above and beyond a behavioral, guideline-based asthma intervention.

To test how well MAST works, a pilot randomized controlled trial (RCT) with 84 urban adolescents (42 = NYC; 42 = RI) with persistent asthma and whose typical sleep duration is at/below what is recommended for this age group. Students will be recruited from high schools in New York City and in Greater Providence, RI, two areas of high asthma prevalence for urban adolescents. Students within schools will be randomized to one of three study arms: (1) MAST -- the new intervention consisting of both asthma and sleep hygiene components; (2) the original ASMA program; and (3) an informational and referral control group. The investigators will follow students for two months post-intervention and explore differences in feasibility, acceptability, and preliminary intervention effects by site.

Following consent, students and their parents/caregivers will complete baseline interviews, and will be randomized into one of the three study conditions. The investigators will deliver the intervention to the students at their respective schools, and will interview students and their parents/caregivers when the intervention ends and two months later. At each assessment, to assess sleep objectively, students will be asked to wear actigraph watches (Model AW2; Mini Mittler) for 2 weeks. During this two week period, they will also complete asthma and sleep logs where they record on a daily basis if they had asthma symptoms, took asthma medication, had asthma-related limitations, and information about their sleep; these logs are completed in the morning and the evening and should take less than 5 minutes each time to complete.

ELIGIBILITY:
Inclusion Criteria: Students will have

* (a) a prior asthma diagnosis;
* (b) used a prescribed asthma medication in the last 12 months; and
* (c) uncontrolled asthma, defined as (i) daytime symptoms 3+ days a week, (ii) night awakenings 3+ nights per month, (iii) 2+ ED visits or (iv) 1+ hospitalization for asthma; and (c) sleep duration 8.5 hours or less (at/below the appropriate number of hours of sleep for this age group through the following questions: What time do you: a) usually fall asleep on weekdays, b) usually wakeup on weekdays?).

Exclusion Criteria:

* report of prior diagnosis of a sleep disorder, such as sleep disordered breathing, restless leg syndrome, periodic limb movement syndrome;
* active immunotherapy;
* additional pulmonary disease; and
* significant developmental delay and/or severe psychiatric or medical conditions that preclude completion of study procedures or confound analyses.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Quality score | Baseline, immediate post-intervention and 2-months post-intervention
  Sleep efficiency will be calculated from data obtain from actigraphs (Model AW2; Mini Mittler) that the teenagers will wear for 2 weeks at each point.

SECONDARY OUTCOMES:
Change in Asthma Control score | Baseline, immediate post-intervention and 2-months post-intervention
  We will use the Asthma Control Test, is a 5-item instrument validated for those 12 and older. Respondents indicate on a five-point scale how often in the past 4 weeks they had symptoms, had activity restrictions, used rescue medication; they also rate their perceived asthma control. Scores range from 5 to 25, with higher scores reflecting greater asthma control. An ACT score of 19 or more indicate well-controlled asthma.. Students will also report using a two-week recall of (a) # of days with symptoms, (b) # of nights woken wakening with symptoms, and (c) how bothered they were by the symptoms. We will also assess symptom severity using Whalgren's asthma symptom scale which rates asthma symptoms during the last 2 weeks on a 5 point scale where 0=none and 4=severe.
Change in Asthma Management Skill - Symptom Prevention Total Score | Baseline, immediate post-intervention and 2-months post-intervention
  We have adapted asthma self-management indices for adolescents developed and used in prior research by our team. These indices assess three categories of management behaviors: (1) symptom prevention; (2) attack management; and (3) self-efficacy in managing asthma. In our middle school study Cronbach's α was 0.67, 0.70, and 0.84 for symptom prevention, attack management, and asthma management self-efficacy, respectively, as reported by students. These scales are treatment sensitive (i.e., detect change in self-care following participation in an intervention). The symptom prevention scale can be used to calculate 2 scores, with one being the Symptom Prevention Total Score ranges from 0 - 27 with higher scores indicating that the teenager takes more steps to prevent symptoms, and does so more regularly.
Change in Asthma Management Skill - Symptom Prevention Steps | Baseline, immediate post-intervention and 2-months post-intervention
  We have adapted asthma self-management indices for adolescents developed and used in prior research by our team. These indices assess three categories of management behaviors: (1) symptom prevention; (2) attack management; and (3) self-efficacy in managing asthma. In our middle school study Cronbach's α was 0.67, 0.70, and 0.84 for symptom prevention, attack management, and asthma management self-efficacy, respectively, as reported by students. These scales are treatment sensitive (i.e., detect change in self-care following participation in an intervention). The symptom prevention scale can be used to calculate 2 scores, with one being the Symptom Prevention Steps ranges from 0 - 9 with higher scores indicating that the teenager takes more steps to prevent the onset of symptoms
Change in Asthma Management Skill - Attack Management score | Baseline, immediate post-intervention and 2-months post-intervention
  We have adapted asthma self-management indices for adolescents developed and used in prior research by our team. These indices assess three categories of management behaviors: (1) symptom prevention; (2) attack management; and (3) self-efficacy in managing asthma. In our middle school study Cronbach's α was 0.67, 0.70, and 0.84 for symptom prevention, attack management, and asthma management self-efficacy, respectively, as reported by students. These scales are treatment sensitive (i.e., detect change in self-care following participation in an intervention). The Attack Management Score ranges from 0 - 7 with higher scores indicating more steps taken to manage existing symptoms
Change in Asthma Management Skill - Self-efficacy Score | Baseline, immediate post-intervention and 2-months post-intervention
  We have adapted asthma self-management indices for adolescents developed and used in prior research by our team. These indices assess three categories of management behaviors: (1) symptom prevention; (2) attack management; and (3) self-efficacy in managing asthma. In our middle school study Cronbach's α was 0.67, 0.70, and 0.84 for symptom prevention, attack management, and asthma management self-efficacy, respectively, as reported by students. These scales are treatment sensitive (i.e., detect change in self-care following participation in an intervention). For the self-efficacy score, the mean of 14 items is calculated with scores ranging from 1 to 6 with higher scores indicated more self-efficacy to care for asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Bruzzese, PhD, Principal Investigator — Columbia University; Daphne Koinis-Mitchell, PhD, Principal Investigator — Rhode Island Hospital
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koinis-Mitchell D, Kopel SJ, Boergers J, McQuaid EL, Esteban CA, Seifer R, Fritz GK, Beltran AJ, Klein RB, LeBourgeois M. Good Sleep Health in Urban Children With Asthma: A Risk and Resilience Approach. J Pediatr Psychol. 2015 Oct;40(9):888-903. doi: 10.1093/jpepsy/jsv046. Epub 2015 May 18. PMID 25991645
- [Background] Vignau J, Bailly D, Duhamel A, Vervaecke P, Beuscart R, Collinet C. Epidemiologic study of sleep quality and troubles in French secondary school adolescents. J Adolesc Health. 1997 Nov;21(5):343-50. doi: 10.1016/S1054-139X(97)00109-2. PMID 9358298
- [Background] Meltzer LJ, Ullrich M, Szefler SJ. Sleep duration, sleep hygiene, and insomnia in adolescents with asthma. J Allergy Clin Immunol Pract. 2014 Sep-Oct;2(5):562-9. doi: 10.1016/j.jaip.2014.02.005. Epub 2014 Apr 13. PMID 25213049
- [Background] Wolfson AR, Carskadon MA. Understanding adolescents' sleep patterns and school performance: a critical appraisal. Sleep Med Rev. 2003 Dec;7(6):491-506. doi: 10.1016/s1087-0792(03)90003-7. PMID 15018092
- [Background] Wolfson AR, Carskadon MA. Sleep schedules and daytime functioning in adolescents. Child Dev. 1998 Aug;69(4):875-87. PMID 9768476
- [Background] Spilsbury JC, Storfer-Isser A, Drotar D, Rosen CL, Kirchner LH, Benham H, Redline S. Sleep behavior in an urban US sample of school-aged children. Arch Pediatr Adolesc Med. 2004 Oct;158(10):988-94. doi: 10.1001/archpedi.158.10.988. PMID 15466688
- [Background] Colrain IM, Baker FC. Changes in sleep as a function of adolescent development. Neuropsychol Rev. 2011 Mar;21(1):5-21. doi: 10.1007/s11065-010-9155-5. Epub 2011 Jan 12. PMID 21225346
- [Background] Dahl RE, Lewin DS. Pathways to adolescent health sleep regulation and behavior. J Adolesc Health. 2002 Dec;31(6 Suppl):175-84. doi: 10.1016/s1054-139x(02)00506-2. PMID 12470913
- [Background] Keyes KM, Maslowsky J, Hamilton A, Schulenberg J. The great sleep recession: changes in sleep duration among US adolescents, 1991-2012. Pediatrics. 2015 Mar;135(3):460-8. doi: 10.1542/peds.2014-2707. PMID 25687142
- [Background] Wong ML, Lau EY, Wan JH, Cheung SF, Hui CH, Mok DS. The interplay between sleep and mood in predicting academic functioning, physical health and psychological health: a longitudinal study. J Psychosom Res. 2013 Apr;74(4):271-7. doi: 10.1016/j.jpsychores.2012.08.014. Epub 2012 Sep 25. PMID 23497826
- [Background] Newacheck PW, Halfon N. Prevalence, impact, and trends in childhood disability due to asthma. Arch Pediatr Adolesc Med. 2000 Mar;154(3):287-93. doi: 10.1001/archpedi.154.3.287. PMID 10710030
- [Background] Worldwide variations in the prevalence of asthma symptoms: the International Study of Asthma and Allergies in Childhood (ISAAC). Eur Respir J. 1998 Aug;12(2):315-35. doi: 10.1183/09031936.98.12020315. PMID 9727780
- [Background] Centers for Disease Control and Prevention (CDC). Self-reported asthma among high school students--United States, 2003. MMWR Morb Mortal Wkly Rep. 2005 Aug 12;54(31):765-7. PMID 16094284
- [Background] Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. Pediatrics. 2009 Mar;123 Suppl 3:S131-45. doi: 10.1542/peds.2008-2233C. PMID 19221156
- [Background] Pearce N, Ait-Khaled N, Beasley R, Mallol J, Keil U, Mitchell E, Robertson C; ISAAC Phase Three Study Group. Worldwide trends in the prevalence of asthma symptoms: phase III of the International Study of Asthma and Allergies in Childhood (ISAAC). Thorax. 2007 Sep;62(9):758-66. doi: 10.1136/thx.2006.070169. Epub 2007 May 15. PMID 17504817
- [Background] Akinbami LJ, Schoendorf KC. Trends in childhood asthma: prevalence, health care utilization, and mortality. Pediatrics. 2002 Aug;110(2 Pt 1):315-22. doi: 10.1542/peds.110.2.315. PMID 12165584
- [Background] Bruzzese JM, Stepney C, Fiorino EK, Bornstein L, Wang J, Petkova E, Evans D. Asthma self-management is sub-optimal in urban Hispanic and African American/black early adolescents with uncontrolled persistent asthma. J Asthma. 2012 Feb;49(1):90-7. doi: 10.3109/02770903.2011.637595. Epub 2011 Dec 7. PMID 22149141
- [Background] Claudio L, Stingone JA, Godbold J. Prevalence of childhood asthma in urban communities: the impact of ethnicity and income. Ann Epidemiol. 2006 May;16(5):332-40. doi: 10.1016/j.annepidem.2005.06.046. Epub 2005 Oct 20. PMID 16242960
- [Background] Koinis-Mitchell D, McQuaid EL, Seifer R, Kopel SJ, Esteban C, Canino G, Garcia-Coll C, Klein R, Fritz GK. Multiple urban and asthma-related risks and their association with asthma morbidity in children. J Pediatr Psychol. 2007 Jun;32(5):582-95. doi: 10.1093/jpepsy/jsl050. Epub 2007 Jan 11. PMID 17218338
- [Background] Wright RJ. Further evidence that the wealthier are healthier: negative life events and asthma-specific quality of life. Thorax. 2007 Feb;62(2):106-8. doi: 10.1136/thx.2006.067926. PMID 17287304
- [Background] Williams DR, Sternthal M, Wright RJ. Social determinants: taking the social context of asthma seriously. Pediatrics. 2009 Mar;123 Suppl 3(Suppl 3):S174-84. doi: 10.1542/peds.2008-2233H. PMID 19221161
- [Background] Clark NM, Brown R, Joseph CL, Anderson EW, Liu M, Valerio M, Gong M. Issues in identifying asthma and estimating prevalence in an urban school population. J Clin Epidemiol. 2002 Sep;55(9):870-81. doi: 10.1016/s0895-4356(02)00451-1. PMID 12393074
- [Background] Koinis-Mitchell D, McQuaid EL, Kopel SJ, Esteban CA, Ortega AN, Seifer R, Garcia-Coll C, Klein R, Cespedes E, Canino G, Fritz GK. Cultural-related, contextual, and asthma-specific risks associated with asthma morbidity in urban children. J Clin Psychol Med Settings. 2010 Mar;17(1):38-48. doi: 10.1007/s10880-009-9178-3. PMID 20157798
- [Background] McLaughlin Crabtree V, Beal Korhonen J, Montgomery-Downs HE, Faye Jones V, O'Brien LM, Gozal D. Cultural influences on the bedtime behaviors of young children. Sleep Med. 2005 Jul;6(4):319-24. doi: 10.1016/j.sleep.2005.02.001. Epub 2005 Apr 1. PMID 15978515
- [Background] Redline S, Tishler PV, Schluchter M, Aylor J, Clark K, Graham G. Risk factors for sleep-disordered breathing in children. Associations with obesity, race, and respiratory problems. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1527-32. doi: 10.1164/ajrccm.159.5.9809079. PMID 10228121
- [Background] Rosen CL, Palermo TM, Larkin EK, Redline S. Health-related quality of life and sleep-disordered breathing in children. Sleep. 2002 Sep 15;25(6):657-66. PMID 12224844
- [Background] Spilsbury JC, Storfer-Isser A, Kirchner HL, Nelson L, Rosen CL, Drotar D, Redline S. Neighborhood disadvantage as a risk factor for pediatric obstructive sleep apnea. J Pediatr. 2006 Sep;149(3):342-7. doi: 10.1016/j.jpeds.2006.04.061. PMID 16939744
- [Background] Boergers J, Koinis-Mitchell D. Sleep and culture in children with medical conditions. J Pediatr Psychol. 2010 Oct;35(9):915-26. doi: 10.1093/jpepsy/jsq016. Epub 2010 Mar 23. PMID 20332222
- [Background] Koinis-Mitchell D, Kopel SJ, Boergers J, Ramos K, LeBourgeois M, McQuaid EL, Esteban CA, Seifer R, Fritz GK, Klein R. Asthma, allergic rhinitis, and sleep problems in urban children. J Clin Sleep Med. 2015 Jan 15;11(2):101-10. doi: 10.5664/jcsm.4450. PMID 25515273
- [Background] Bruzzese JM, Bonner S, Vincent EJ, Sheares BJ, Mellins RB, Levison MJ, Wiesemann S, Du Y, Zimmerman BJ, Evans D. Asthma education: the adolescent experience. Patient Educ Couns. 2004 Dec;55(3):396-406. doi: 10.1016/j.pec.2003.04.009. PMID 15582346
- [Background] Bruzzese JM, Sheares BJ, Vincent EJ, Du Y, Sadeghi H, Levison MJ, Mellins RB, Evans D. Effects of a school-based intervention for urban adolescents with asthma. A controlled trial. Am J Respir Crit Care Med. 2011 Apr 15;183(8):998-1006. doi: 10.1164/rccm.201003-0429OC. Epub 2010 Dec 7. PMID 21139088